CLINICAL TRIAL: NCT05553496
Title: Assessment of Rituximab Therapeutic Response Versus Conventional Treatment in the Management of Refractory Nephrotic Syndrome
Brief Title: Assessment of Rituximab Therapeutic Response Versus Conventional Treatment
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, shaymaa omar, Head of clinical pharmacy department at Dar Al Fouad hospital, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHCL555
Record Dates: First submitted 2022-09-15; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Pharmacological Action
MeSH Terms: interventions — Rituximab; Dexamethasone; Tacrolimus; Cyclophosphamide; Cyclosporine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RTX in Refractory Nephrotic syndrome patients on conventional treatment (Active Comparator): Refratory Nephrotic syndrome participants will receive a 375 mg/m2 weekly rituximab for four doses, with retreatment every 2 months till 6 months regardless of proteinuria response in addition to triple optimized immunosuppression therapy including steroids ± Calcineurine inhibitors (CNI) (e.g: Tacrolimus), Mycophenloatemofetil (MMF) and Cyclophosphamide (CTX)
  Interventions: Drug: Rituximab; Drug: Dexamethasone
- Refractory Nephrotic Syndrome patients on Conventional therapy (Active Comparator): Nephrotic syndrome participants will receive conventional therapy treatment only including steroids ± Tacrolimus (TAC), Cyclosporine (CsA), Mycophenloatemofetil (MMF), and Cyclophosphamide (CTX) then if become refractory to conventional treatment will continue on the same treatment.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Rituximab — Group (1) RTX in Refractory Nephrotic syndrome patients on conventional treatment (20 patients)
  Other Names: Dexamethasone; Tacrolimus; Mycophenloatemofetil; Cyclophosphamide
  Arms: RTX in Refractory Nephrotic syndrome patients on conventional treatment
Drug: Dexamethasone — Group (2) Refractory Nephrotic Syndrome patients on Conventional therapy (20 patients)
  Other Names: Tacrolimus; Cyclosporine; Mycophenloatemofetil; Cyclophosphamide

SUMMARY:
Prospective interventional comparative study to compare the efficacy of Rituximab versus Conventional treatment in Refractory Nephrotic Syndrome including patients on triple immunosuppression protocols.

DETAILED DESCRIPTION:
A prospective randomized controlled interventional study, conducted on Refractory Nephrotic syndrome patients with failed different lines of conventional treatment.

The aim of the current study is to assess the therapeutic response of Rituximab versus Conventional treatment in Refractory Nephrotic Syndrome in terms of :

* Improvement in proteinuria.
* Relapse frequency.

Fourty patients with Refractory Nephrotic syndrome will be enrolled in the study. All participants will be previously treated with ACEi and/or ARB, for ≥3 months prior to randomization and adequate blood pressure control. Participants will be assigned randomly into two groups with 20 Refractory Nephrotic syndrome patients in each group as follow:

* Group (1) RTX in Refractory Nephrotic syndrome patients on conventional treatment (20 patients)
* Group (2) Refractory Nephrotic Syndrome patients on Conventional therapy (20 patients)

The duration and severity of proteinuria are known to be surrogate markers of the progression of glomerular disease. Our approach to assess the clinical response was to evaluate estimated Glomerular filtration rate (eGFR), proteinuria and serum albumin after rituximab treatment. We classified the response into four stages :

1. No proteinuria, normal serum albumin
2. Mild proteinuria, serum albumin >30 g/l
3. Ongoing significant proteinuria, serum albumin 20-30 g/l
4. No change in proteinuria and serum albumin. Stages 1 and 2 will be interpreted as a good clinical response, whereas stages 3 and 4 will be interpreted as a poor clinical response.

A sample size of fourty patients with Refractory Nephrotic syndrome is selected to achieve confidence limit of 5%. At the end of the study, a number of data will be generated, such as:

1. Quantitative data will be summarized as means and standard deviations and/or medians and ranges.
2. Categorical data will be summarized as frequencies & percentage.
3. For measuring statistical differences between groups, categorical variables are analyzed using the chi-squared test or Fisher's exact test, whereas continuous variables are compared using Student t tests or Mann-Whitney U tests or Wilcoxon signed-rank test, as appropriate.
4. Statistical comparisons between pre- and post-treatment values are performed using the Wilcoxon signed-rank test.
5. Univariate linear regression models are used to examine the association between baseline characteristics and response to drug treatment.
6. All tests are performed at a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 year old and medically stable.
2. Treatment with an Angiotension converting enzyme inhibitor (ACEi) and/or Angiotension II receptor blockade (ARB), for ≥3 months prior to randomization and adequate blood pressure control or if patient is intolerant to even a very low dose of either ACEi or ARB therapy.
3. Proteinuria ≥3 g/24 h using the average from two 24-hour urine collections collected within 14 days of each other despite ARB for ≥3 months as described above.
4. Estimated GFR ≥40 ml/min/1.73 m2 while taking ACEi/ARB therapy or quantified endogenous creatinine clearance ≥40 ml/min based on a 24 h urine collection.
5. Non responsive GN patients on conventional treatment.

Exclusion Criteria:

1. Autoimmune diseases.
2. Patients with presence of active infection or a secondary cause of IMN (e.g. hepatitis B, SLE, medications, malignancies).
3. Type 1 or 2 diabetes mellitus: to exclude proteinuria secondary to diabetic nephropathy.
4. Pregnancy or breast feeding.
5. Predisposition to drug hypersensitivity.
6. Unstable medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-25 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of either conventional therapy alone or Rituximab as an add on therapy will be assessed by measure of Remission sate of the patient. | 6 months
  The primary end point is Complete or Partial remission at 6 months after randomization. Complete remission (CR) is defined as UP ≤0.3 g/24 h and serum albumin ≥3.5 g/dl while Partial remission (PR) is defined as Reduction in baseline UP of ≥50% plus final UP ≤3.5 g/24 h but >0.3 g/24 h. The patient who will be Non-responsive to therapy is defined as Reduction in baseline UP of <25% (includes increase in UP) after 6 months of immunosuppression and the patient who will enter in the relapsed phase is defined as development of nephrotic range proteinuria following CR or PR, i.e. >3.5 g/24 h.

SECONDARY OUTCOMES:
A) Late Remissions: | 6, 9, and 12 months after randomization.
  The first 6 months of the study will be considered the treatment period, while the remaining 6 months will be considered an observational period.So we will monitor the patients for CR or PR at 6, 9, and 12 months after randomization.
B) Relapse state: | 12 months after randomization
  Relapse state of the patient will be assessed at month 12 after randomization (Urine Protein (UP) >3.5 g/24 h after earlier CR or PR).
C) Response Treatment Time: | 12 months after randomization
  The response time will be assessed by measuring the duration of clinical response to RTX in patients who had on going CR or PR.
D) End Stage Renal Disease (ESRD): | 12 months after randomization
  The patients who developed ESRD will be reviewed in this study.
E) Renal Function: | 6 months after randomization
  The effect of treatment on renal function will be assessed every 3 months by calculating the estimated GFR (eGFR) with the creatinine-based Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula from baseline to 6 months.
F) Adverse events: | 6, 9, and 12 months after randomization.
  Patients will be educated about adverse effects of the drugs and will be required to report the occurrence of any of them.